CLINICAL TRIAL: NCT03453346
Title: Evaluation of Safety and Efficacy of Generic Sofosbuvir and Ribavirin for Treatment-naive Adults Chronically Infected With Genotype 2 Hepatitis C Virus: an Open-label, Multicenter Confirmatory Study
Brief Title: Safety and Efficacy of Generic Sofosbuvir and Ribavirin for Treatment-naive Genotype 2 Chronic Hepatitis C
Acronym: SOF_GT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kawin Technology Share-holding Co., Ltd. (Industry)
Collaborators: KawinGreen Biotech Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJKY-2016-003; CTR20160399 (Registry Identifier: China Drug Trials)
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Hepatitis C, Chronic; Hepatitis C Virus Infection, Response to Therapy of
Keywords: Hepatitis C virus; Sofosbuvir; RNA polymerase inhibitor; Ribavirin; Genotype 2; Sustained virologic response; Confirmatory study
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Sofosbuvir; Ribavirin

STUDY DESIGN:
Intervention Model Description: Open label, single arm, historical control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Noncirrhotic and cirrhotic GT-2 (Experimental): Generic sofosbuvir tablet 400 mg once daily plus weight-adjusted ribavirin tablet (1000 mg for <75 kg, and 1200 mg for >=75 kg) twice daily with meal, orally given, for 12 successive weeks
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir — Generic sofosbuvir tablet 400 mg
  Other Names: SOF
Drug: Ribavirin — Ribavirin was provided in 100-mg tablets.
  Other Names: RBV

SUMMARY:
This study aimed to evaluate the safety and efficacy of generic sofosbuvir, an investigational anti-hepatitis C virus (HCV) drug, combined with weight-adjusted ribavirin for treatment-naive Chinese adults chronically infected with genotype 2 HCV, the second most prevalent genotype in China. One hundred and thirty-two (132) subjects, including one hundred and twenty (120) non-cirrhotics and twelve (12) compensatory cirrhotics, were medicated with sofosbuvir 400 mg daily combined with weight-adjusted ribavirin 1000-1200 mg daily. The treatment course lasted 12 successive weeks and thereafter all the study participants entered into a 12-week treatment-free follow-up period.

DETAILED DESCRIPTION:
It is estimated that China has a population of over 10 million infected with HCV and also a highly variable HCV genotype geographic distribution. Genotype 2 HCV is reported to be the second most common type (~25%) in Chinese population and associated with a high risk of acute liver disease exacerbation and other extrahepatic diseases. Sofosbuvir is a pan-genotypic HCV ribonucleic acid (RNA) polymerase inhibitor directing at HCV RNA replication. Genotype 2 chronic hepatitis C has a high treatment response to the combined regimen of peginterferon and weight-adjusted ribavirin. The all-oral combination regimen of sofosbuvir and ribavirin is expected to completely suppress genotype 2 HCV replication in subjects chronically infected with HCV and achieve a sustained virologic response, namely, HCV not detected or below a predefined limit in plasma, 12 or 24 weeks after cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years (inclusive) and of either sex
* with a body mass index (BMI) between 18 and 30 kg/m^2
* chronically infected with genotype 2 HCV, and the diagnosis of chronic hepatitis C consistent with the Chinese Guideline for Prevention and Management of Hepatitis C
* HCV RNA equaling to or above 10^4 IU/mL and anti-HCV positivity
* naive to anti-HCV treatment, defined as being not previously treated with any interferon (including interferon alfa or beta or peginterferon), ribavirin, or other approved, investigational or any other not approved anti-HCV regimens of any source
* with or without cirrhosis, presence or absence of which must be documented as at lease one item of the following: 1) liver biopsy confirming presence (e.g., Metavir score = 4 or Ishak score >=5) or absence of cirrhosis within twelve (12) months before screening; 2) FibroScan showing cirrhosis (liver stiffness modulus [LSM]>=12.5 kPa) or no cirrhosis (LSM=<9.6 kPa); 3) a subject with a LSM of 9.6-12.5 kPa (exclusive) could only be enrolled when the liver biopsy confirmed or excluded presence of cirrhosis
* women of childbearing potential without a history of menopause and with a negative blood pregnancy test; subjects of childbearing potential (including male subjects and their female partners) had no childbearing plan from screening, initiation of treatment until six (6) months after the end of treatment and consented to use effective contraceptive measures
* voluntary participation in the study and being able to understand and sign the informed consent form

Exclusion Criteria:

* being infected with mixed-genotype HCV
* having previously used any investigational or experimental direct antiviral agents against HCV, including protease, nonstructural (NS) protein 5B polymerase or NS5A inhibitors, before screening
* having received any interferon-based anti-HCV regimens before screening
* having been exposed to any systemic potent immunomodulators , such as steroids or thymosin alfa (excluding use of nasal, inhalational, topical steroids and/or others) for more than two (2) weeks within six (6) months before screening, or anticipated to be exposed to these agents during the study period
* being coinfected with hepatitis B virus (HBV) or human immunodeficient virus (HIV)
* with evidence of decompensatory liver function, including but not limited to total serum bilirubin (TBIL) above twice (2) of the upper limit of normal (ULN), serum albumin (ALB) below 35 g/L, or prothrombin activity (PTA) below 60%; emergence of ascites, upper gastrointestinal bleeding and/or hepatic encephalopathy; with liver function reserve Child-Pugh class B or C
* with primary liver cancer confirmed or evidenced by serum alfa-fetoprotein above 100 ng/ml or liver imaging study showing suspected nodules
* with a previous history of liver disease of other causes, including alcoholic liver disease, nonalcoholic steatohepatitis, drug-induced hepatitis, autoimmune hepatitis (anti-nuclear antibody[ANA] titer above 1:100), Wilson disease or hemochromatosis
* with serum alaine aminotransferase (ALT) or asparate aminotransferase (AST) above ten (10) times of ULN
* with white blood cell (WBC) count below 3x10^9 per liter, neutrophil count below 1.5x10^9 per liter, platelet count below 50x10^9 per liter, or hemoglobin below the lower limit of the normal
* with serum creatinine clearance (CLcr) below 50 ml/min using the Cockcroft-Gault formula
* with uncontrolled diabetes mellitus (hemoglobin A1c[HbA1c] above 7.0%)
* with psychiatric or neurologic disorders, including previous or family history of psychiatric disorders (especially depression, depressive state, epilepsy or hysteria)
* with serious cardiovascular disorders, including uncontrolled hypertension (systolic blood pressure at or above 160 mmHg and/or diastolic blood pressure at or above 100 mmHg), heart insufficiency of New York Heart Association class III or above, history of myocardial infarction within six (6) months before screening, history of percutaneous transluminal coronary angioplasty within six (6) months before screening, unstable angina pectoris, or any uncontrolled arrhythmias
* with serious hematologic disorders (such as anemia, hemophilia and others)
* with serious kidney diseases (such as chronic kidney disease, kidney insufficiency and others)
* with serious gastrointestinal disorders (such as peptic ulcer, colitis and others)
* with serious respirator disorders (such as active pulmonary tuberculosis, lung infection, chronic obstructive pulmonary disease, pulmonary interstitial disease and others)
* with active or suspected malignant tumors or with a previous history of malignant tumors (excluding skin basal cell carcinoma or cervical carcinoma in situ) within five (5) years before screening
* with a history of major organ transplantation
* being known to be severely hypersensitive or allergic to any drugs, especially the testing medications and other constituents
* with a history of active alcohol or drug abuse
* being pregnant or lactating
* being unable to discontinue prohibited medications as defined by the protocol
* having participated in any other clinical studies within three (3) months before screening
* being unable or unwilling to provide informed consent or unable to follow the protocol requirements
* any other conditions of excluding a potential participant at the discretion of the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2017-03-18 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response at 12 weeks after end of treatment (SVR12) | 12 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)

SECONDARY OUTCOMES:
Sustained virologic response at 4 weeks after end of treatment (SVR4) | 4 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 1 week after initiation of treatment (RVR1) | 1 week after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 2 weeks after initiation of treatment (RVR2) | 2 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 4 weeks after initiation of treatment (RVR4) | 4 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 8 weeks after initiation of treatment (RVR8) | 8 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 12 weeks after initiation of treatment (RVR12) | 12 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)

OTHER OUTCOMES:
Virologic breakthrough | 2, 4, 8 and 12 weeks after initiation of treatment
  Percentage of subjects with on-treatment re-detected plasma HCV RNA after HCV RNA below the lower limit of quantitation
Virologic relapse | 4 and 12 weeks after end of treatment
  Percentage of subjects with off-treatment re-detected plasma HCV RNA after end-of-treatment HCV RNA below the lower limit of quantitation

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, M.D., Principal Investigator — Peking University People's Hospital
Locations (17):
- China (17):
  - Chinese PLA 302 Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing Youyi Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing You'an Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Chongqing Medical University Affiliated Second Hospital, Chongqing, Chongqing Municipality
  - Chinese PLA Third Military Medical University First Affiliated Hospital, Chongqing, Chongqing Municipality
  - He'nan Provincial People's Hospital, Zhengzhou, He'nan
  - He'nan Provincial Hospital of Infectious Disease (Zhengzhou Municipal Sixth People's Hospital), Zhengzhou, He'nan
  - Hebei Medical University Affiliated Third Hospital, Shijiazhuang, Hebei
  - Nanjing Municipal Second Hospital, Nanjing, Jiangsu
  - Jilin University First Hospital, Changchun, Jilin
  - Shenyang Municipal Sixth People's Hospital, Shenyang, Liaoning
  - Chinese PLA Fourth Military Medical University Tangdu Hospital, Xi'an, Shaanxi
  - Xi'an Jiaotong University College of Medicine Affiliated First Hospital, Xi'an, Shaanxi
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan was included in the study protocol.